CLINICAL TRIAL: NCT05271942
Title: Tilt and Tumble vs Divide and Conquer - a Unique Comparison of the Two Cataract Surgery Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aleris Eye (Industry)
Responsible Party: Principal Investigator, Johan Ursberg, Chief Medical Officer, Aleris Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aleris Eye
Record Dates: First submitted 2021-09-15; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Cataract
Keywords: Divide and Conquer, Tilt and Tumble
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Randomization into two groups
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tilt and Tumble (Experimental): The patients of this group will undergo cataract surgery using the "Tilt and Tumble" technique.
  Interventions: Procedure: Tilt and Tumble
- Divide and Conquer (Active Comparator): The patients of this group will undergo cataract surgery using the "Divide and Conquer" technique.
  Interventions: Procedure: Divide and Conquer

INTERVENTIONS:
Procedure: Tilt and Tumble — The Tilt and Tumble technique is used to remove the human lens.
  Arms: Tilt and Tumble
Procedure: Divide and Conquer — The Divide and Conquer technique is used to remove the human lens.
  Arms: Divide and Conquer

SUMMARY:
The purpose of this study is to compare two different methods used during cataract surgery to remove the lens in the eye.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants who have signed the written informed consent will be randomized to undergo cataract surgery with either the method called "Divide and Conquer" or "Tilt and Tumble". Pre- per- and postoperative measurements from the surgery will be filed and compared later on by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Cataract

Exclusion Criteria:

* Dementia
* Very narrow anterior chamber
* Born after 1965

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Differences in energy during phacoemulsification between the methods investigated. | Immediately after the surgery
  Energy used during phacoemulsification is measured during each surgery. It is measured with the unit Cumulative Dissipated Energy (CDE).
Differences in time used during phacoemulsification during surgery between the methods investigated | Immediately after the intervention/procedure/surgery
  Time, measured in seconds (s), will be measured from the start til the end of phacoemulsification
Difference in corneal endothelial cell density after cataract surgery between the study groups investigated. Before and after surgery. Change is being assessed. | Pre-intervention surgery and 14 days after surgery.
  During cataract surgery the participants loose some of the endothelial cells. The investigator can measure endothelial cell density (CD) with an endothelial cell camera. This will be done before and after surgery in both study groups.
Measurement of clinical och subclinical macular oedema before and after surgery. Change is being assessed. | Pre-intervention surgery and 14 days after surgery.
  Clinical or subclinical macular oedema is a known complication to cataract surgery. Macula will be measured with an Ocular Coherence Tomography (OCT) before and after surgery. Retinal thickness in macula will be measured in micrometer. Data is collected after each surgery from the phaco apparatus throughout the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Aleris Eye Clinci, Helsingborg, Skåne County
  - Aleris Eye Clinic, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 2023